CLINICAL TRIAL: NCT06313437
Title: A Phase I Trial of Revumenib in Combination With 7+3 (7 Days of Cytarabine and 3 Days of Daunorubicin) + Midostaurin Induction Chemotherapy for the Frontline Treatment of NPM1 and FLT3 Mutated AML
Brief Title: Revumenib in Combination With 7+3 + Midostaurin in AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Stone, MD (Other)
Collaborators: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Richard Stone, MD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-021
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia; AML, Adult; AML With Gene Mutations; AML; Leukemia
Keywords: Acute Myeloid Leukemia; AML, Adult; AML with Gene Mutations; AML; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — revumenib; midostaurin; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Revumenib (Experimental): Standard 3+3 design for a recommended phase 2 dose of Revumenib per dose-limiting toxicity rules. Cycles are 28 days.
  * Baseline
  * Induction Cycle:
    * Days 1-3: Predetermined dose of Daunorubicin 1x daily
    * Days 1-7: Predetermined dose of Cytarabine
    * Days 8-21: Predetermined dose of Midostaurin 2x daily
    * Days 8-28: Predetermined dose of Revumenib 2x daily
  * End of Induction visit
  * Follow-up
  * Reinduction Cycle: Therapy will be administered in the hospital
    * Days 1-2: Predetermined dose of Daunorubicin 1x daily
    * Days 1-5: Predetermined dose of Cytarabine
    * Days 8-21: Predetermined dose of Midostaurin 2x daily
    * Days 8-28: Predetermined dose of Revumenib 2x daily
  * End of reinduction visit
  * Follow-up
  * Consolidation Cycle: Therapy will be administered in the hospital
    * Days 1, 3, and 5: Predetermined dose of Cytarabine
    * Days 8-21: Predetermined dose of Midostaurin 2x daily
    * Days 8-28: Predetermined dose of Revumenib 2x daily
  * End of consolidation visit
  * Follow up
  Interventions: Drug: Revumenib; Drug: Midostaurin; Drug: Cytarabine; Drug: Daunorubicin
- Dose-Expansion Revumenib (Experimental): Cycles are 28 days
  * Baseline visit and assessments
  * Induction Cycle:
    * Days 1-3: Predetermined dose of Daunorubicin 1x daily
    * Days 1-7: Predetermined dose of Cytarabine
    * Days 8-21: Predetermined dose of Midostaurin 2x daily
    * Days 8-28: Predetermined dose of Revumenib 2x daily
  * End of Induction visit
  * Follow-up
  * Reinduction Cycle: Therapy will be administered in the hospital
    * Days 1-2: Predetermined dose of Daunorubicin 1x daily
    * Days 1-5: Predetermined dose of Cytarabine
    * Days 8-21: Predetermined dose of Midostaurin 2x daily
    * Days 8-28: Predetermined dose of Revumenib 2x daily
  * End of Reinduction visit
  * Follow-up
  * Consolidation Cycle: Therapy will be administered in the hospital
    * Days 1, 3, and 5: Predetermined dose of Cytarabine
    * Days 8-21: Predetermined dose of Midostaurin 2x daily
    * Days 8-28: Predetermined dose of Revumenib 2x daily
  * End of Consolidation visit
  * Follow up
  Interventions: Drug: Revumenib; Drug: Midostaurin; Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: Revumenib — Menin inhibitor, 25 and 113 mg capsules, taken orally per protocol.
  Other Names: SNDX-5613; Trans N-ethyl-2-((4-(7-((4-(ethylsulfonamido)cyclohexyl)methyl)-2,7-diazaspiro[3.5]nonan-2- yl)pyrimidin-5-yl)oxy)-5-fluoro-N-isopropylbenzamide
Drug: Midostaurin — Kinase inhibitor, capsule taken orally per protocol.
  Other Names: Rydapt
Drug: Cytarabine — Antineoplastic agent, via intravenous (into the vein) infusion per protocol.
  Other Names: cytosine arabinoside (ara-C)
Drug: Daunorubicin — Antineoplastic agent, via intravenous (into the vein) infusion per protocol.
  Other Names: Daunomycin

SUMMARY:
This research is being conducted to determine a safe and effective dose of revumenib that can be given in combination with standard induction (initial therapy to induce a remission) + FLT3 targeted therapy (midostaurin) and a single cycle of post-remission therapy + FLT3 targeted therapy (midostaurin) to participants with newly diagnosed Nucleophosmin (NPM1) and FMS-like tyrosine kinase 3 (FLT3) mutated Acute Myeloid Leukemia (AML).

The names of the study drugs involved in this study are:

* Revumenib (SNDX-5613) (a type of menin inhibitor)
* Midostaurin (a type of multi-kinase including FLT3 inhibitor)
* Cytarabine (a type of antineoplastic agent)
* Daunorubicin (a type of antineoplastic agent)

DETAILED DESCRIPTION:
This is a single arm open label phase I trial of the menin inhibitor, revumenib, in combination with cytarabine and daunorubicin (7+3) chemotherapy and the multikinase inhibitor midostaurin for the frontline treatment of Nucleophosmin (NPM1) and FMS-like tyrosine kinase 3 (FLT3) mutated Acute Myeloid Leukemia (AML).

Investigators are trying to determine the highest dose of revumenib that can be given safely in combination with these chemotherapy drugs. Treatment consists of 1-2 cycles of so-called "induction treatment" (initial chemotherapy to induce a remission of the leukemia). This "induction treatment" consists of revumenib + 7+3 (7 days of cytarabine + 3 days of daunorubicin) chemotherapy + midostaurin.

The U.S. Food and Drug Administration (FDA) has not approved the combination of revumenib, cytarabine, daunorubicin, and midostaurin as a treatment for AML.

The research study procedures include screening for eligibility, study treatment visits, blood and urine tests, bone marrow biopsies, and electrocardiograms (ECGs).

Participants will receive study treatment as long as there are no serious side effects and the disease does not progress.

The trial will include up to 12 participants in dose finding phase and 10 additional participants in the dose expansion phase for a total participant number of 22 participants.

Syndax Pharmaceuticals is supporting this research study by supply revumenib (SNDX-5613).

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML who are newly diagnosed according to the WHO 2022 Classification and previously untreated except for hydroxyurea. ATRA pretreatment for suspected APL for less than 5 days is allowed. Eligible patients with AML arising from an antecedent hematologic disease (AHD) including MDS, may have been treated for their prior hematologic disease (except for allogenic transplant).
* Patients must be ≥ 18 and < 75 years old.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 2.
* Presence of FLT3-ITD and/or TKD mutation(s) AND NPM1 mutation in bone marrow or peripheral blood
* Dose escalation phase only: Presence of any of the following adverse risk genetic characteristics:

  * 2022 ELN adverse risk genetic features:

    * t(6;9)(p23.3;q34.1)/DEK::NUP214
    * t(v;11q23.3)/KMT2A-rearranged
    * t(9;22)(q34.1;q11.2)/BCR::ABL1
    * t(8;16)(p11.2;p13.3)/KAT6A::CREBBP
    * inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2)/ GATA2, MECOM(EVI1)
    * t(3q26.2;v)/MECOM(EVI1)-rearranged
    * -5 or del(5q); -7; -17/abn(17p)
    * Complex karyotype, monosomal karyotype
    * Mutations in either one of these genes: ASXL1, BCOR, EZH2, RUNX1, SF3B1, SRSF2, STAG2, U2AF1, and/or ZRSR2
    * Mutated TP53
  * NPM1 + FLT3-ITD + DNMT3A mutation
* LVEF ≥ 50% by MUGA or ECHO at screening.
* Adequate renal function as demonstrated by a calculated creatinine clearance ≥ 60 mL/min; determined by the Cockcroft Gault formula.
* Adequate liver function as demonstrated by:

  * aspartate aminotransferase (AST) ≤ 2.5 × ULN*
  * alanine aminotransferase (ALT) ≤ 2.5× ULN*
  * total bilirubin ≤ 1.5 × ULN* * Unless considered due to leukemic organ involvement. Note: Subjects with Gilbert's Syndrome may have a total bilirubin > 1.5 × ULN per discussion with the Sponsor-Investigator
* Resolution of adverse reactions to prior drug therapy (such as hydroxyurea) to ≤ grade 1
* Eligible for intensive cytarabine/daunorubicin (7+3) chemotherapy based on the opinion of the treating physician.
* Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 90 days after the last dose of study drug.
* Females of childbearing potential (i.e., not postmenopausal for at least 1 year or not surgically sterile) must have negative results by a serum or urine pregnancy test performed within 7 days of day 1.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)
* Consolidation should occur between 1-4 weeks following count recovery after induction and remission (must be confirmed by labs to document maximal response) is established. Subjects will receive medium intensity cytarabine -based consolidation in combination with midostaurin and revumenib if the following criteria are fulfilled.

  * an induction response < 5% blasts in the bone marrow and ANC >1000 and PLT >75000 for whom documented path report is submitted.
  * sufficiently fit (performance status <3)
  * resolution of any adverse reactions to no greater than grade 1 severity

Exclusion Criteria:

* Subject has acute promyelocytic leukemia, inversion (16), t(8;21) AML as described below. Contact Sponsor-Investigator with questions. Inversion 16 and t(8;21): CBF chromosomal abnormalities may be assessed by molecular (PCR), metaphase cytogenetics, or FISH.
* Subject has known active CNS involvement with AML.
* Subject has received a strong CYP3A4 inducer (APPENDIX C) within 7 days prior to the initiation of study treatment
* Strong CYP3A4 inhibitors (APPENDIX C) are contraindicated except strong CYP3A4 inhibitor antifungal azole medications (systemic itraconazole, ketoconazole, posaconazole, voriconazole). For strong CYP3A4 inhibitor antifungal azole medications, the starting dose of revumenib has to be adjusted (Table 1).
* QTc using Fridericia's correction [QTcF]) > 450 msec. Drugs that prolong QTc should be avoided if possible. A list of common QTc prolonging drugs and alternatives that are not QTc prolonging can be found in APPENDIX D.
* Subject has tested positive for HIV (due to potential drug-drug interaction between antiretroviral medications and Midostaurin/revumenib). Note: HIV testing is not required.
* Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load within 3 months. (Hepatitis B or C testing is not required). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and antiHBs+] are allowed.
* Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit within 3 days prior to the initiation of study treatment.
* Subject has a cardiovascular disability status of New York Heart Association Class ≥ 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
* Subject has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study.
* Subject has chronic respiratory disease that requires continuous oxygen use.
* Subject has a malabsorption syndrome or other condition that precludes enteral route of administration.
* Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to uncontrolled systemic infection.
* Subject has a history of other malignancies prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
  * Prior malignancies treated with (surgery+/- chemotherapy+/- radiation) that have remained disease free for at least two years after completion of therapy
* Subject treated with any form of chemotherapy, immunotherapy, or investigative agent within 1 month of enrollment.
* Patients who have had prior exposure to a menin inhibitor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose Limiting Toxicity (DLT) | Up to 12 weeks
  Detailed DLT consideration outline in protocol section 5.4.
Maximum Tolerated Dose (MTD) | Up to 12 weeks
  MTD is determined by the number of patients who experience a DLT. See previous primary outcome measure for the DLT definition. If 0 out of 3 participants experience DLT, next dose level will be proceeded. If >=1 out of the group suffer DLT, dose escalation will be stopped and 3 additional participants will be entered at the next lowest dose level. If <=1 out of 6 DLTs, this dose level is considered as MTD.
Recommended phase II dose (RP2D) | Up to 12 weeks
  The RP2D is determined by a combination of the MTD (see previous primary outcome measure), pharmacokinetics, pharmacodynamics and response rate to different doses of revumenib in combination with chemotherapy and the FLT3 inhibitor midostaurin.

SECONDARY OUTCOMES:
Complete Remission (CR) rate with induction chemotherapy | Up to 8 weeks
  CR rate is defined as the proportion of participants who achieve a CR as defined by the ELN 2022 response criteria after completion of induction chemotherapy.
Complete Remission (CR) rate with consolidation chemotherapy | Up to 12 weeks
  CR rate is defined as the proportion of participants who achieve a CR as defined by the ELN 2022 response criteria after completion of consolidation chemotherapy.
Flow Measurable Residual Disease Negative (MRD-) rate with induction chemotherapy | Up to 8 weeks
  Flow MRD rate is defined as the proportion of participants who achieve MRD negativity (MRD-) after completion of induction chemotherapy assessed by MRD sensitive flow cytometry.
Flow Measurable Residual Disease Negative (MRD-) rate with consolidation chemotherapy | Up to 12 weeks
  Flow MRD rate is defined as the proportion of participants who achieve MRD negativity (MRD-) after completion of consolidation chemotherapy assessed by MRD sensitive flow cytometry.
Molecular Measurable Residual Disease Negative (MRD-) rate with induction chemotherapy | Up to 8 weeks
  Molecular MRD rate is defined as the proportion of participants who achieve MRD negativity (MRD-) after completion of induction chemotherapy as assessed by NPM1 MRD testing as well as FLT3 ITD MRD testing and duplex sequencing.
Molecular Measurable Residual Disease Negative (MRD-) rate with consolidation chemotherapy | Up to 12 weeks
  Molecular MRD rate is defined as the proportion of participants who achieve MRD negativity (MRD-) after completion of consolidation chemotherapy as assessed by NPM1 MRD testing as well as FLT3 ITD MRD testing and duplex sequencing.
Relapse-Free Survival at 1 year (RFS1) | Up to 1 year
  RFS is defined as the length of time after the completion of a particular medical treatment during which a patient remains free of any signs or symptoms of disease relapse or recurrence based on Kaplan-Meier methodology.
Overall Survival at 1 year (OS1) | Up to 1 year
  OS1 is the probability estimated using the Kaplan-Meier method; OS is defined as the time from study entry to death, or censored at the date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu